CLINICAL TRIAL: NCT03066180
Title: Pilot Study of Non-Ablative Radiofrequency Treatment for Stress Urinary Incontinence
Brief Title: Study of Non-Ablative Radiofrequency Treatment for Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Bruce B. Allan (Other)
Responsible Party: Sponsor-Investigator, Dr. Bruce B. Allan, Bruce B. Allan, PhD, MD, FRCSC, Allan Centre
Organization: Allan Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VI-ERP-010
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 (Experimental): Single study treatment (Viveve SUI treatment) will be administered.
  Interventions: Device: Viveve SUI treatment
- Group 2 (Experimental): Two study treatments (Viveve SUI treatments) will be administered approximately 6 weeks apart.
  Interventions: Device: Viveve SUI treatment

INTERVENTIONS:
Device: Viveve SUI treatment — Non-ablative radiofrequency treatment with surface cooling

SUMMARY:
This is a prospective, pilot clinical study involving two study groups. This study is designed to demonstrate that the study treatment meets primary efficacy and safety endpoints. The treatment involves radiofrequency treatment to address symptoms of stress urinary incontinence.

After receiving the study treatment, subjects will be followed out to 12 months post-treatment. At the Screening Visit, and at each designated follow-up timepoint, subjects will be asked to complete a variety of questionnaires, provide a patient diary, and undergo an objective assessment for urine loss.

DETAILED DESCRIPTION:
This is a prospective, pilot clinical study involving two study groups. Subjects meeting the all the inclusion criteria and none of the exclusion criteria will be enrolled in the study. Subjects will receive a single SUI treatment; subjects in Group 2 will receive two SUI Treatments.

At the Screening Visit, and at each pre-designated study follow-up timepoint, subjects will be asked to complete several quality of life questionnaires related to the treated condition. In addition, subjects will provide a bladder voiding diary for review and data collection, and a pad weight test will be conducted and results collected.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and has voluntarily signed and dated the informed consent form (ICF) prior to initiation of any screening or study-specific procedures.
* Willing to comply with study requirements and instructions.
* Female, ≥ 18 years of age.
* Normal pelvic exam at Screening.
* Negative pregnancy test at Screening.
* Diagnosed with mild or moderate Stress Urinary Incontinence (SUI) by the 1-hour pad weight test ("mild" defined as 1 - 10 g; "moderate" defined as 11 - 50 g; and "severe" defined as >50 g ) at Screening.

Exclusion Criteria:

* Subject is currently breastfeeding or discontinued breast feeding fewer than 6 months prior to enrollment.
* Any condition, illness, or surgery that might confound the results of urinary incontinence assessment, including, but not limited to:

  * Categories of urinary incontinence other than the categories being investigated.
  * Prominent (i.e., greater than stage II as defined by the International Continence Society) pelvic organ prolapse (e.g., cystocele, rectocele).
  * Neurological disorders (e.g., multiple sclerosis, Parkinson's disease).
  * Spastic bladder.
  * Concurrent infections (e.g., urinary tract infection [UTI], cystitis, urethritis, active genital herpes flare-up, active genital/pelvic infection).
  * Vesicoureteral reflux.
  * Bladder stones.
  * Bladder tumors.
  * Morbid obesity.
* Any underlying condition that may pose unreasonable risks to the subject, such as:

  * Coagulation abnormalities.
  * Abnormal kidney function.
  * Uncontrolled diabetes.
  * Has an implantable electrical device [e.g., implantable pacemaker, automatic implantable cardioverter-defibrillator (AICD)] that could potentially be affected by the use of radiofrequency.
* Taking any new medication (< 3 months) that affects urination, or change in the dosage of any medication that affects urination within the past 3 months.
* Medical history of keloid formation, genital fistula, thin recto-vaginal septum (defined as a distance of < 2 cm between the vaginal opening and the anal opening, as measured by a flexible tape measure); or history of fourth-degree laceration, hypertrophic scar formation, or mediolateral episiotomy.
* Active malignancy or undergoing treatment (using chemotherapeutic agents, radiation therapy, and/or cytostatic medications) that may interfere with adequate wound healing response.
* Previous vaginal, energy-based device treatment for vaginal laxity, urinary incontinence, or sexual function (e.g., radiofrequency treatment, cosmetic, laser, surgical, and/or genital enhancement procedure).
* Chronic use of anti-inflammatory drugs, including ibuprofen, aspirin, and steroids.
* Subject has been in another clinical study within 6 months of screening, or is not willing to abstain from participating in other clinical studies for duration of trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
reduction in pad weight vs. baseline | baseline to 12 months post-treatment
  pad weight tests to be completed at baseline and at designated study follow-up timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Bruce B Allan, PhD, MD, Principal Investigator — University of Calgary
Locations (1):
- Allan Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Shumaker SA, Wyman JF, Uebersax JS, McClish D, Fantl JA. Health-related quality of life measures for women with urinary incontinence: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res. 1994 Oct;3(5):291-306. doi: 10.1007/BF00451721. PMID 7841963
- [Background] Harvey MA, Kristjansson B, Griffith D, Versi E. The Incontinence Impact Questionnaire and the Urogenital Distress Inventory: a revisit of their validity in women without a urodynamic diagnosis. Am J Obstet Gynecol. 2001 Jul;185(1):25-31. doi: 10.1067/mob.2001.116369. PMID 11483899
- [Derived] Allan BB, Bell S, Husarek K. Early Feasibility Study to Evaluate the Viveve System for Female Stress Urinary Incontinence: Interim 6-Month Report. J Womens Health (Larchmt). 2020 Mar;29(3):383-389. doi: 10.1089/jwh.2018.7567. Epub 2019 Aug 29. PMID 31464548